CLINICAL TRIAL: NCT04164199
Title: An Open-Label, Multicenter, Long-Term Extension Study of Treatment With Tislelizumab, Pamiparib, and Other Investigational Agents in Patients With Advanced Malignancies
Brief Title: Study of Tislelizumab, Pamiparib, and Other Investigational Agents in Participants With Advanced Malignancies
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-290-LTE1; 2019-002554-23 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — tislelizumab; pamiparib; Temozolomide; sitravatinib; HMPL-013; zanidatamab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- A - Tislelizumab Monotherapy (Experimental)
  Interventions: Drug: Tislelizumab
- B - Pamiparib Monotherapy (Experimental)
  Interventions: Drug: Pamiparib
- C - Sitravatinib Monotherapy (Experimental)
  Interventions: Drug: Sitravatinib
- D - BGB-15025 Monotherapy (Experimental)
  Interventions: Drug: BGB-15025
- E - Zanidatamab Monotherapy (Experimental)
  Interventions: Drug: Zanidatamab
- F - Pamiparib and Temozolomide Combination Therapy (Experimental)
  Interventions: Drug: Pamiparib; Drug: Temozolomide
- G - Tislelizumab and Pamiparib Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Pamiparib
- H - Tislelizumab and Sitravatinib Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Sitravatinib
- I - Tislelizumab and Ociperlimab Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Ociperlimab
- J - Tislelizumab and BAT1706 Combination Therapy, or BAT1706 Monotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: BAT1706
- K - Tislelizumab and Fruquintinib Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib
- L - Tislelizumab and BGB-A445 Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: BGB-A445
- M - Tislelizumab and Surzebiclimab Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Surzebiclimab
- N - Tislelizumab and BGB-15025 Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: BGB-15025
- O - Tislelizumab and Lenvatinib Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Lenvatinib
- P - Tislelizumab and Zanidatamab Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Zanidatamab
- Q - Tislelizumab and LBL-007 Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: LBL-007
- R - Tislelizumab and Surzebiclimab and LBL-007 Combination Therapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Surzebiclimab; Drug: LBL-007

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously.
  Other Names: BGB-A317
  Arms: A - Tislelizumab Monotherapy; G - Tislelizumab and Pamiparib Combination Therapy; H - Tislelizumab and Sitravatinib Combination Therapy; I - Tislelizumab and Ociperlimab Combination Therapy; J - Tislelizumab and BAT1706 Combination Therapy, or BAT1706 Monotherapy; K - Tislelizumab and Fruquintinib Combination Therapy; L - Tislelizumab and BGB-A445 Combination Therapy; M - Tislelizumab and Surzebiclimab Combination Therapy; N - Tislelizumab and BGB-15025 Combination Therapy; O - Tislelizumab and Lenvatinib Combination Therapy; P - Tislelizumab and Zanidatamab Combination Therapy; Q - Tislelizumab and LBL-007 Combination Therapy; R - Tislelizumab and Surzebiclimab and LBL-007 Combination Therapy
Drug: Pamiparib — Administered orally.
  Other Names: BGB-290
  Arms: B - Pamiparib Monotherapy; F - Pamiparib and Temozolomide Combination Therapy; G - Tislelizumab and Pamiparib Combination Therapy
Drug: Temozolomide — Administered orally.
  Arms: F - Pamiparib and Temozolomide Combination Therapy
Drug: Sitravatinib — Administered orally.
  Arms: C - Sitravatinib Monotherapy; H - Tislelizumab and Sitravatinib Combination Therapy
Drug: Ociperlimab — Administered intravenously.
  Other Names: BGB-A1217
  Arms: I - Tislelizumab and Ociperlimab Combination Therapy
Drug: BAT1706 — Administered intravenously.
  Arms: J - Tislelizumab and BAT1706 Combination Therapy, or BAT1706 Monotherapy
Drug: Fruquintinib — Administered orally.
  Arms: K - Tislelizumab and Fruquintinib Combination Therapy
Drug: BGB-15025 — Administered orally.
  Arms: D - BGB-15025 Monotherapy; N - Tislelizumab and BGB-15025 Combination Therapy
Drug: Zanidatamab — Administered intravenously.
  Other Names: ZW25
  Arms: E - Zanidatamab Monotherapy; P - Tislelizumab and Zanidatamab Combination Therapy
Drug: BGB-A445 — Administered intravenously.
  Other Names: Gimistotug
  Arms: L - Tislelizumab and BGB-A445 Combination Therapy
Drug: Surzebiclimab — Administered intravenously.
  Other Names: BGB-A425
  Arms: M - Tislelizumab and Surzebiclimab Combination Therapy; R - Tislelizumab and Surzebiclimab and LBL-007 Combination Therapy
Drug: Lenvatinib — Administered orally.
  Arms: O - Tislelizumab and Lenvatinib Combination Therapy
Drug: LBL-007 — Administered intravenously.
  Other Names: Alcestobart
  Arms: Q - Tislelizumab and LBL-007 Combination Therapy; R - Tislelizumab and Surzebiclimab and LBL-007 Combination Therapy

SUMMARY:
This is an open-label, multicenter, extension study to evaluate the long-term safety and efficacy of BeiGene investigational drugs in participants with advanced malignancies who participated in a prior BeiGene-sponsored clinical study (parent study).

DETAILED DESCRIPTION:
For the purposes of this study, "study treatment" will refer to all investigational agents. A parent study is defined as the original BeiGene-sponsored clinical trial in which the participant was initially enrolled and received BeiGene investigational drugs (with or without other treatments).

ELIGIBILITY:
Key Inclusion Criteria:

1. Currently participating in a BeiGene-sponsored eligible parent study
2. Fulfills treatment criteria specified in the parent study protocol
3. In the opinion of the investigator, the participant will continue to benefit from and tolerate any of the parent study treatments.
4. The first dose of study treatment in the LTE study will be received within the treatment interruption period allowed by the parent study:

   1. "Treatment interruption" (unplanned pause in study treatment) and "treatment break" (planned stop of study therapy) are not interchangeable. Restarting study treatment beyond the interruption period allowed by the parent study or after a treatment break will be determined by the investigator and the sponsor. Participants who have not restarted treatment within 1 year of starting a treatment break must discontinue treatment.

Specific Inclusion Criteria for Participants Who Continue Survival Follow-up Only in the Extension Study:

1. Currently participating in a BeiGene-sponsored eligible parent study in the survival follow-up portion
2. Parent study plans to have survival analysis

Key Exclusion Criteria:

1. Permanently discontinued from all investigational drugs in the parent study due to unacceptable toxicity, noncompliance with study procedures, or withdrawal of consent
2. Have uncontrolled active systemic infection or recent infection requiring parenteral antimicrobial therapy prior to the start of the extension study
3. Have a life-threatening illness, medical condition, or organ system dysfunction that in the investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of investigational drugs, or put the study outcomes at undue risk
4. Underwent treatment with any systemic anticancer treatment (other than treatment permitted in the parent study) during the time between the last treatment in the parent study and the first dose of study treatment in the LTE study
5. Pregnant or lactating women

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Immune-Mediated Adverse Events | up to 7 years
  Safety as assessed by the number of participants with immune-mediated adverse events related to immunotherapy as assessed by the investigator, > Grade 3 adverse events, Grade 2 adverse events that affect key organs (eg, heart, liver, brain, lung, kidney, eye), nonserious adverse events that lead to dose modification or drug discontinuation or withdrawal from the trial, and serious adverse events.

SECONDARY OUTCOMES:
Overall survival | up to 7 years
  Overall survival defined as the time from start of treatment in the parent study (or randomization date for a randomized parent study) until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (106):
- United States (4):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
- Australia (7):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- China (50):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital Sun Yat Sen University, Zhuhai, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Affiliated Hospital of Zunyi Medical University, Zuiyi, Guizhou
  - Hainan Cancer Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University Wuhan, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Provincial Wenzhou Hospital of Zhejiang, Wenzhou, Zhejiang
- France (5):
  - Hopital Beaujon, Clichy
  - Hopital Prive Jean Mermoz, Lyon
  - Icm Val Daurelle, Montpellier
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Larchet Chu Nice, Nice
- Italy (3):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Aou Pisana, Stabilimento Di Santa Chiara, Pisa
  - Azienda Ospedaliera S Maria Di Terni, Terni
- Japan (7):
  - Akita University Hospital, Akitashi, Akita
  - Chiba Cancer Center, Chiba, Chiba
  - Nho Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Izumi City General Hospital, Izumishi, Osaka
  - The University of Osaka Hospital, Suitashi, Osaka
  - National Cancer Center Hospital, ChuoKu, Tokyo
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Auckland City Hospital, Auckland, New Zealand
- Poland (2):
  - Szpitale Pomorskie Spolka Z Ograniczona Odpowiedzialnoscia, Gdynia
  - Centrum Onkologii Instytut Im M Sklodowskiej Curie, Warsaw
- South Korea (14):
  - Cha Bundang Medical Center, Cha University, BundangGu SeongnamSi, Gyeonggi-do
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, PaldalGu SuwonSi, Gyeonggi-do
  - Gachon University Gil Medical Center, NamdongGu, Incheon Gwang'yeogsi
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Smg Snu Boramae Medical Center, DongjakGu, Seoul Teugbyeolsi
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Korea University Guro Hospital, GuroGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
  - Ajou University Hospital, Suwon
- Taiwan (7):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Linkou Chang Gung Memorial Hospital, Guishan Dist
  - Kaohsiung Chang Gung Memorial Hospital, Niaosong Dist
  - China Medical University Hospital, North Dist
  - National Cheng Kung University Hospital, North Dist
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Yongkang Dist
- King Chulalongkorn Memorial Hospital (Chulalongkorn University), Pathum Wan, Thailand
- Turkey (Türkiye) (3):
  - Acibadem Adana Hospital, Kuruköprü
  - Bakirkoy Sadi Konuk Eah, stanbulBakrkoy
  - Namik Kemal University, Tekirdağ

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/